CLINICAL TRIAL: NCT05610475
Title: Serum Level of Calpains Product as a Novel Biomarker of Acute Lung Injury Following Cardiopulmonary Bypass(CPB)
Brief Title: Serum Level of Calpains Product as a Novel Biomarker of Acute Lung Injury Following Cardiopulmonary Bypass
Acronym: CPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 20220201
Record Dates: First submitted 2022-10-30; First posted 2022-11-09 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Lung Injury, Acute
Keywords: Cardiopulmonary Bypass; Calpain; Lung injury
MeSH Terms: conditions — Acute Lung Injury; Lung Injury | interventions — Echocardiography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung injury group (Active Comparator)
  Interventions: Diagnostic Test: blood cell analysis, blood gas surveillance, chest radiograph and echocardiography
- Non-lung injury group (Sham Comparator)
  Interventions: Diagnostic Test: blood cell analysis, blood gas surveillance, chest radiograph and echocardiography

INTERVENTIONS:
Diagnostic Test: blood cell analysis, blood gas surveillance, chest radiograph and echocardiography — Laboratory parameters of all postoperative patients including blood cell analysis, blood gas surveillance, liver, and kidney function alone with chest radiograph and echocardiography were dynamically monitored.

SUMMARY:
More than 2 million patients worldwide receive heart surgery every year, majority of these surgical patients will undergo cardiopulmonary bypass. However, the incidence of postoperative acute lung injury due to cardiopulmonary bypass is still as high as 20% to 35%. According to clinical experience, the earlier lung damage is detected, the more successful the treatment will be. On the basis of traditional detection, the investigators found a new indicator, serum calpains, which are easy to obtain and have certain specificity. Importantly, they can predict postoperative acute lung injury within 1 hour after cardiac surgery. It is meaningful that this indicator can provide clinicians with early decision-making advice and immediate treatment for patients who may be at risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Underwent cardiac surgery using CPB technology.

Exclusion criteria :

* Patient's lack of consent to participate;
* Presence of abnormal liver, kidney or other organ function;
* Pulmonary inflammation, chronic obstructive pulmonary disease or tumors;
* Underwent cardiac surgery without CPB technology;
* Postoperative need for extracorporeal membrane oxygenation support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | Change from beginning of CPB to 48 h after CPB
  The ratio of inspiratory oxygen fraction to oxygen pressure (PaO2/FiO2) was calculated.
lung-injury scores | The 24 and 48 hours after CPB
  A structured tutorial was used to establish consensus in the interpretation of radiographs for radiographic lung-injury scores, range from 0 to 4.
  0: No alveolar consolidation; 1: Alveolar consolidation confined to 1 quadrant; 2: Alveolar consolidation confined to 2 quadrants 3: Alveolar consolidation confined to 3 quadrants; 4: Alveolar consolidation in all 4 quadrants.
  The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Perioperative serum calpains' concentrations | The day before CPB and 1, 12, 24, 48 hours after CPB
  Serial serum samples were obtained and measured by using a fluorometric kit (Abcam, Cambridge, UK) according to the manufacturer's protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China

REFERENCES:
- [Derived] Yi C, Chen F, Ma R, Fu Z, Song M, Zhang Z, Chen L, Tang X, Lu P, Li B, Zhang Q, Song Q, Zhu G, Wang W, Wang Q, Wang X. Serum level of calpains product as a novel biomarker of acute lung injury following cardiopulmonary bypass. Front Cardiovasc Med. 2022 Nov 16;9:1000761. doi: 10.3389/fcvm.2022.1000761. eCollection 2022. PMID 36465445